CLINICAL TRIAL: NCT02420652
Title: A Phase 2 Randomized Discontinuation Trial in Patients With Hormone-Dependent Rising Prostate-Specific Antigen Progression After Local Therapy for Prostate Cancer Evaluating the Synergy of Metformin Plus Aspirin (PRIMA Trial)
Brief Title: Metformin Hydrochloride and Aspirin in Treating Patients With Hormone-Dependent Prostate Cancer That Has Progressed After Surgery or Radiation Therapy
Acronym: PRIMA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Principal Investigator, Biren Saraiya, MD, Assistant Professor of Medicine, Rutgers Cancer Institute of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 081501; NCI-2015-00397 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro20150001378 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Recurrent Prostate Carcinoma; Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Aspirin; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (metformin hydrochloride, aspirin) (Experimental): Patients receive metformin hydrochloride PO BID and aspirin PO QD for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Aspirin; Other: Laboratory Biomarker Analysis; Drug: Metformin Hydrochloride
- Arm II (metformin hydrochloride placebo, aspirin placebo) (Placebo Comparator): Patients receive metformin hydrochloride placebo PO BID and aspirin placebo PO QD for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo

INTERVENTIONS:
Drug: Aspirin — Given PO
  Other Names: Acetylsalicylic Acid; ASA; Aspergum; Ecotrin; Empirin; Entericin; Extren; Measurin
  Arms: Arm I (metformin hydrochloride, aspirin)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Metformin Hydrochloride — Given PO
  Other Names: Glucophage; Metformin HCl
  Arms: Arm I (metformin hydrochloride, aspirin)
Other: Placebo — Given metformin hydrochloride placebo PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (metformin hydrochloride placebo, aspirin placebo)
Other: Placebo — Given aspirin placebo PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (metformin hydrochloride placebo, aspirin placebo)

SUMMARY:
This randomized phase II trial studies how well metformin hydrochloride and aspirin work in treating patients with hormone-dependent prostate cancer that has progressed after surgery or radiation therapy. Metformin hydrochloride and aspirin may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether giving metformin hydrochloride and aspirin together can slow the growth of prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effect of metformin (metformin hydrochloride) and aspirin on the change in prostate-specific antigen (PSA) progression in men with rising PSA after definitive therapy for localized prostate cancer and stable disease during a run-in period with the study regimen.

SECONDARY OBJECTIVES:

I. To determine the feasibility and safety of administering metformin and aspirin.

II. To determine the effect of metformin and aspirin on PSA levels and the serum obesity-related prostate cancer (PCa) biomarkers (insulin, insulin-like growth factor [IGF]-1, interleukin [IL]-1beta, IL-6, and tumor necrosis factor [TNF]-alpha).

OUTLINE:

RUN-IN STAGE: Patients receive metformin hydrochloride orally (PO) twice daily (BID) and aspirin PO once daily (QD) for 4 months. Patients with disease progression (PSA increase of > 50% and minimum of 2ng/ml rise in PSA) come off study. Patients achieving disease response (>25% decline in PSA) continue to receive study agents in the absence of disease progression or unacceptable disease. Patients with stable disease continue on to the randomized study regimen.

RANDOMIZATION STAGE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive metformin hydrochloride PO BID and aspirin PO QD for 6 months in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive metformin hydrochloride placebo PO BID and aspirin placebo PO QD for 6 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12-16 weeks for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven prostate cancer treated with surgery, radiation, or the combination of surgery and radiation for prostate cancer (metastatic to regional lymph nodes) with resection of the nodes, who now has a rising PSA value after definitive local therapy, and no visible metastatic disease on conventional imaging studies
* Patients must have undergone local treatment via prostatectomy or radiation therapy
* Patients must have PSA progression after local treatment:

  * PSA values for patients after surgery (or surgery and salvage/adjuvant radiation) must be greater than or equal to 0.2 ng/mL, determined by two measurements, at least 1 month apart and at least 6 months after prostatectomy
  * PSA values for patients after radiation must be greater than or equal to 2.0 ng/ml greater than the nadir achieved after radiation, determined by two measurements at 1 month apart and at least 6 months after the radiation treatment is completed; (patients who received adjuvant or salvage radiation after prostatectomy must have PSA of greater than or equal to 0.2)
  * The first two PSA values, along with a third (study baseline) value must all be rising (i.e., there must be an overall rising trajectory, such that the third value cannot be lower than the first value)
  * PSA must be less than 50 ng/mL at study entry
  * PSA doubling time using the mkscc.org PSA doubling time calculator must be greater than 4 months
* Baseline bone scan, chest x-ray and computed tomography (CT)/magnetic resonance imaging (MRI) of abdomen/pelvis demonstrating no metastatic disease
* Estimated life expectancy of at least 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* White blood cells (WBC) > 3500/ul
* Absolute neutrophil count (ANC) > 1500/ul
* Hemoglobin > 10 g/dl
* Platelet count > 100,000/ul
* Adequate renal function with estimated glomerular filtration rate (GFR) by Cockcroft Gault of greater than 40 ML per minute
* Total bilirubin must be within 1.5 X the normal institutional limits; if total bilirubin is outside the normal institutional limits, assess direct bilirubin
* The direct bilirubin must be within normal parameters
* Transaminases (serum glutamic oxaloacetic transaminase [SGOT] and/or serum glutamate pyruvate transaminase [SGPT]) must be less than 2.5 X the institutional upper limit of normal
* Patients must have a serum total testosterone level >= 150 ng/dL at the time of enrollment within 4 weeks prior to randomization
* Patients must sign informed consent

Exclusion Criteria:

* Serious concomitant systemic disorder that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator
* Patients may have received prior androgen deprivation therapy (ADT) in the neoadjuvant, adjuvant and/or salvage setting, but must be off therapy for at least 3 months and have a testosterone level > 150 ng/dl
* Second primary malignancy except most situ carcinoma (e.g. adequately treated non-melanomatous carcinoma of the skin) or other malignancy treated at least 2 years previously with no evidence of recurrence
* Patients with type II diabetes currently already on metformin
* Patients taking aspirin for previously diagnosed cardiovascular disease
* Patients who received aspirin or metformin within the past 28 days
* Patients taking medications with known interactions with metformin or aspirin
* Patients taking warfarin or platelet inhibitors
* Patients requiring chronic use of nonsteroidal anti-inflammatory drugs (NSAIDS)
* Other concurrent experimental or investigational drugs
* Prior history of lactic acidosis or metabolic acidosis
* Patients with history of gastrointestinal (GI) bleeding and peptic ulcer disease
* Any unstable, serious co-existing medical conditions including but not limited to myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias, clinically evident congestive heart failure, or cerebrovascular accident within 6 months prior to screening

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-06-23 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Biren Saraiya, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Metformin Hydrochloride, Aspirin) | Arm II (Metformin Hydrochloride Placebo, Aspirin Placebo)
Started | 18 | 9
Completed | 8 | 5
Not Completed | 10 | 4

BASELINE CHARACTERISTICS:
Groups:
- Arm I (Metformin Hydrochloride, Aspirin): Patients receive metformin hydrochloride placebo PO BID and aspirin placebo PO QD for 6 months in the absence of disease progression or unacceptable toxicity.
- Arm II (Metformin Hydrochloride Placebo, Aspirin Placebo): Metformin 1500 mg/Day and Aspirin 81 mg/Day x 4 cycles. Participants receive metformin hydrochloride PO BID and aspirin PO QD for 6 months in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Arm I (Metformin Hydrochloride, Aspirin) | Arm II (Metformin Hydrochloride Placebo, Aspirin Placebo) | Total
Number analyzed (Participants) | 18 | 9 | 27
Age, Continuous [Mean (Full Range); unit: years] | 67.8 [53 to 83] | 67.8 [53 to 83] | 67.8 [53 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 18 | 9 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 17 | 8 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: Measure of PSA ng/mL Rates After Six Months of Metformin Hydrochloride and Aspirin or Placebo Therapy in Patients Who Have Received Four Months of Open Label Treatment
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm I (Metformin Hydrochloride, Aspirin) | Arm II (Metformin Hydrochloride Placebo, Aspirin Placebo)
Number analyzed (Participants) | 8 | 5
ng/mL | 2.02 (0.77) | 1.43 (0.54)

ADVERSE EVENTS:
Time Frame: Adverse events data was collected up to one year
Arm/Group | Arm I (Metformin Hydrochloride, Aspirin) | Arm II (Metformin Hydrochloride Placebo, Aspirin Placebo)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/5
Other Adverse Events (participants affected / at risk) | 0/8 | 0/5

LIMITATIONS AND CAVEATS:
Early termination lead to a small number of study participants being analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT02420652/Prot_SAP_000.pdf
  • Informed Consent Form (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT02420652/ICF_001.pdf